CLINICAL TRIAL: NCT01644123
Title: Inter-Rater Reliability of a Spasticity Diagnosis Algorithm
Brief Title: Reliability of an Algorithm to Diagnose Spasticity
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, David Charles, Vice-Chairman, Department of Neurology; Chief Medical Officer, Vanderbilt Neuroscience Institute, Vanderbilt University
Other Study IDs: 090361; 090361 (Other: Vanderbilt IRB)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Spasticity
Keywords: Spasticity; Diagnostic Algorithm
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nursing home residents

SUMMARY:
Spasticity is a condition that results from damage to the central nervous system and causes painful muscle contractures that drastically affect level of independence, activities of daily living, and quality of life. Although there are well-known and accepted treatments for spasticity, spasticity is often left undertreated; the specific reasons for this observation are unknown. Because there is no blood test or scan that indicates the presence of spasticity, diagnosis is based entirely on physician impression. Therefore, the investigators hypothesize that one reason that spasticity is undertreated is due to the lack of a standardized diagnostic procedure. This study attempts to test the reliability of a diagnostic flowchart that seeks to increase the accuracy of physician diagnosis of spasticity.

DETAILED DESCRIPTION:
Spasticity is defined as a velocity-dependent increase in stretch reflex with muscle overactivity, and is associated with involuntary limb movements or spasms which can often be painful. Active function (such as walking, driving, writing, or sexual activity) can be adversely affected by spasticity. For patients with significant disability requiring a caregiver, passive function (such as facilitation of bathing, dressing, and undergarment change) can also become very difficult, especially when spasticity is left untreated. Finally, persistent involuntary motion or spasms may negatively impact an individual's mood or self image, making social situations more difficult and sometimes overwhelming.

Spasticity is especially undertreated in vulnerable populations; population surveys in individuals with intellectual disability and nursing home residents have shown that less than 20% of affected individuals are treated. There are severe negative consequences of leaving spasticity untreated, like muscle shortening and tendon and soft tissue contractures. Once developed, contractures are very difficult to treat and can hinder personal hygiene and dressing, and well as the ability to sit or lie properly. Bad hygiene and immobility can lead, in turn, to urinary tract infections, pressure ulcers and skin breakdown. Furthermore, spasticity can stunt muscle growth and cause abnormal bone growth and formation, especially in children.

Spasticity is diagnosed based upon a physician's clinical impression; there is currently no biomarker to facilitate an objective diagnosis. The two instruments most commonly used to document severity are the Modified Ashworth Scale and Range of Motion Assessment. Both assessments are based upon a clinician's assessment of muscle tone, but there is no widely-accepted protocol to determine the presence of spasticity. We therefore hypothesize one reason spasticity is widely undertreated is the challenge faced by physicians when attempting to make a diagnosis. In the absence of a biomarker, a more standardized method of clinical diagnosis is necessary, both for future research and for advocacy efforts. The treatment of spasticity could increase quality of life by allowing an individual to participate more independently in activities of daily living, and by making assistance easier for caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any race, aged 18 and above.
* Reside in one of the five selected long term care facilities.

Exclusion Criteria:

* Subjects for whom it is felt that participation in the study would cause medical harm.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability of a spasticity diagnosis algorithm when used by two movement disorder specialists. | One year
  Two movement disorders specialists will independently use the flowchart while performing physical and neurological examinations on enrolled patients to determine whether spasticity is present.

SECONDARY OUTCOMES:
To compare the prevalence of spasticity between three nursing homes in Davidson County, Tennessee. | One year
  We will attempt to estimate the prevalence of spasticity in the nursing home setting based on the prevalence observed in 3 randomly selected nursing homes in Middle Tennessee.
Awareness of different spasticity treatments and treatment preferences (if treatment is applicable) based on a Treatment Preferences Survey. | One year
  We will survey enrolled subjects to determine if they are aware of available treatments for spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, M.D., Principal Investigator — Vanderbilt University Medical Center; Thomas Davis, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Tennessee State Veterans Home, Murfreesboro, Tennessee
  - Trevecca Health & Rehab, Nashville, Tennessee
  - Bethany Health & Rehabilitation Center, Nashville, Tennessee

REFERENCES:
- [Background] Charles PD, Gill CE, Taylor HM, Putman MS, Blair CR, Roberts AG, Ayers GD, Konrad PE. Spasticity treatment facilitates direct care delivery for adults with profound intellectual disability. Mov Disord. 2010 Mar 15;25(4):466-73. doi: 10.1002/mds.22995. PMID 20131401
- [Background] Gill CE, Andrade EO, Blair CR, Taylor HM, Charles D. Combined treatment with BTX-A and ITB for spasticity: case report. Tenn Med. 2007 Oct;100(10):41-2, 44. PMID 17966716
- [Background] Pfister AA, Roberts AG, Taylor HM, Noel-Spaudling S, Damian MM, Charles PD. Spasticity in adults living in a developmental center. Arch Phys Med Rehabil. 2003 Dec;84(12):1808-12. doi: 10.1016/s0003-9993(03)00368-x. PMID 14669188